CLINICAL TRIAL: NCT05459883
Title: Hemodynamic Modulations to Ameliorate Sinusoidal Injuries After Extended Liver Resections: the Role of Splenic Artery Ligation and Porto-caval Shunt in a Series of Patients
Brief Title: Splenic Artery Ligation and Portocaval Shunt in Small-for-size Syndrome
Acronym: splen ligation
Status: Completed | Type: Observational
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Other Study IDs: 418/18-04-2022
Record Dates: First submitted 2022-07-10; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Small-For-Size Liver Syndrome; Ligation; Liver Regeneration; Splenic Artery; Portal Vein; Ischemia; Reperfusion Injury; Hepatectomy
Keywords: small-for-size liver syndrome; ligation; splenic artery; hepatectomy; liver regeneration
MeSH Terms: conditions — Ischemia; Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: splenic artery ligation — We identified portal hyperperfusion as a cause of potential small-for-size liver remnant dysfunction and we applied splenic artery ligation as a technically simple procedure to manage the situation

SUMMARY:
Our study aimed at assessing the changes of portal vein pressure, portal vein flow and hepatic arterial flow (HAF) in liver remnants ≤ 30% of the standard liver volume by reducing portal vein overflow via ligation of the splenic artery.

DETAILED DESCRIPTION:
It has been reported that prevention of acute portal overpressure in small-for-size liver grafts leads to better postoperative outcomes. Accordingly, we aimed to investigate the feasibility of the technique of splenic artery ligation in a case series of patients subjected to major liver resections with evidence of small-for-size syndrome and whether the maneuver results in reduction of portal venous pressure and flow.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* American Society of Anesthesiologists (ASA) distribution I to III
* Patients scheduled for major liver resection (≥4 segments)

Exclusion Criteria:

* patients with extrahepatic disease
* patients with metastatic liver tumors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: retrospective analysis of an internal hepatectomy database
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
portal vein pressure | through the operation, an average period of two hours
  change of portal vein pressure from before liver resection to after reperfusion of the liver remnant
portal vein flow | through the operation, an average period of two hours
  change of portal vein flow from before liver resection to after reperfusion of the liver remnant
hepatic artery flow | through the operation, an average period of two hours
  change of hepatic artery flow from before liver resection to after reperfusion of the liver remnant

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, Principal Investigator — Aretaieion University Hospital, Athens, Greece
Locations (1):
- Aretaieion University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Theodoraki K, Arkadopoulos N, Nastos C, Vassiliou I, Karmaniolou I, Smyrniotis V. Small liver remnants are more vulnerable to ischemia/reperfusion injury after extended hepatectomies: a case-control study. World J Surg. 2012 Dec;36(12):2895-900. doi: 10.1007/s00268-012-1779-6. PMID 22956015
- [Background] Garcia-Valdecasas JC, Fuster J, Charco R, Bombuy E, Fondevila C, Ferrer J, Ayuso C, Taura P. Changes in portal vein flow after adult living-donor liver transplantation: does it influence postoperative liver function? Liver Transpl. 2003 Jun;9(6):564-9. doi: 10.1053/jlts.2003.50069. PMID 12783396
- [Background] Kinaci E, Kayaalp C. Portosystemic Shunts for "Too Small-for-Size Syndrome" After Liver Transplantation: A Systematic Review. World J Surg. 2016 Aug;40(8):1932-40. doi: 10.1007/s00268-016-3518-x. PMID 27160453
- [Background] Lo CM, Liu CL, Fan ST. Portal hyperperfusion injury as the cause of primary nonfunction in a small-for-size liver graft-successful treatment with splenic artery ligation. Liver Transpl. 2003 Jun;9(6):626-8. doi: 10.1053/jlts.2003.50081. PMID 12783407
- [Background] Umeda Y, Yagi T, Sadamori H, Matsukawa H, Matsuda H, Shinoura S, Mizuno K, Yoshida R, Iwamoto T, Satoh D, Tanaka N. Effects of prophylactic splenic artery modulation on portal overperfusion and liver regeneration in small-for-size graft. Transplantation. 2008 Sep 15;86(5):673-80. doi: 10.1097/TP.0b013e318181e02d. PMID 18791439